CLINICAL TRIAL: NCT00901147
Title: An Open-label Phase 2 Study of Intravenous Bortezomib and Oral Panobinostat (LBH589) in Adult Patients With Relapsed/Refractory Peripheral T-cell Lymphoma or NK/T-cell Lymphoma After Failure of Conventional Chemotherapy
Brief Title: Study of Bortezomib and Panobinostat in Treating Patients With Relapsed/Refractory Peripheral T-cell Lymphoma or NK/T-cell Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Singapore General Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SGH651; SHF/CTG023/2008
Record Dates: First submitted 2009-05-11; First posted 2009-05-13 (Estimated); Last update posted 2014-06-27 (Estimated); Status verified 2014-06

CONDITIONS: Peripheral T-cell Lymphoma (Not Otherwise Specified); Angioimmunoblastic T-cell Lymphoma; Extranodal NK/T-cell Lymphoma Nasal Type; Enteropathy- Type T-cell Lymphoma; Hepatosplenic T-cell Lymphoma; Anaplastic Large Cell Lymphoma (ALCL) (ALK-1 Negative); Relapsed ALCL (ALK-1 Positive) Post Autologous Transplant
Keywords: t-cell lymphoma; peripheral t-cell lymphoma; nk/t-cell lymphoma, nasal type; bortezomib; velcade; panobinostat; LBH589b; histone deacetylase inhibitor; proteasome inhibitor
MeSH Terms: conditions — Lymphoma, T-Cell; Immunoblastic Lymphadenopathy; Lymphoma, Extranodal NK-T-Cell; Enteropathy-Associated T-Cell Lymphoma; Lymphoma, Large-Cell, Anaplastic; Lymphoma, T-Cell, Peripheral | interventions — Panobinostat; Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- panobinostat and bortezomib (Experimental): Oral Panobinostat and intravenous bortezomib
  Interventions: Drug: panobinostat and bortezomib

INTERVENTIONS:
Drug: panobinostat and bortezomib — oral panobinostat 30 mg 3 times per week AND intravenous bortezomib 1.3mg/m2 on days 1,4,8,11 per cycle
  Other Names: LBH589B; Velcade

SUMMARY:
The purpose of this study is to determine whether intravenous Bortezomib combined with oral Panobinostat (LBH589) are effective in treating adult patients with relapsed/refractory peripheral T-cell lymphoma or NK/T-cell lymphoma after the failure of conventional chemotherapy.

DETAILED DESCRIPTION:
Peripheral T-cell lymphoma (PTCL) and NK/T-cell lymphoma are uncommon diseases that are prevalent in Asia. They are associated with poor prognosis when treated with conventional chemotherapeutic regimes. Their long term disease-free survivals are dismal with only 10-30% of patients surviving long term. More intensive regimens including high dose chemotherapy with autologous stem cell transplant have been tried as primary induction treatment, but have not been shown to be beneficial. Given the rarity of PTCL and NK/T-cell lymphoma, much of the literature consists of studies with small sample size and anecdotal case reports. Therefore, no consensus exists on the best therapeutic strategy for either newly diagnosed or relapsed disease. The failure of conventional chemotherapy in this regard suggests that novel therapies including epigenetic approaches and proteasome inhibition should be explored.

Preclinical data of bortezomib and histone deacetylase inhibitors (HDIs) in T-cell and NK/T-cell lymphoma cell lines are encouraging. Bortezomib and HDIs have also separately demonstrated activity in T and NK/T-cell lymphomas in phase II studies, leading to their separate developments in phase III studies. Demonstration of synergism in these 2 agents, in part due to their dependence on overlapping pathways, suggests that they should be explored as a combination, especially when treating a disease with a very unfavourable outcome. The purpose of this phase II study is to assess the efficacy of orally-administered panobinostat, a potent class I/II pan-deacetylase inhibitor with intravenous bortezomib in this patient population.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed PTCL NOS, angioimmunoblastic T-cell lymphoma, extranodal NK/T-cell lymphoma nasal type, enteropathy- type T-cell lymphoma, hepatosplenic T-cell lymphoma, ALCL (ALK-1 negative), or patients with ALK 1 expressing ALCL (ALK-1 positive) who have relapsed disease after ASCT
* Age ≥21 years
* Written informed consent
* Progressive disease following at least one systemic therapy or refractory to at least one prior systemic therapy
* Measurable disease according to the IWC criteria and/or measurable bone marrow disease by flow cytometry or morphology
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Absolute neutrophil count of ≥1000 × 10(9)cells/L
* Serum potassium ≥3.8 mmol/L and magnesium ≥0.85 mmol/L (electrolyte abnormalities can be corrected with supplementation to meet inclusion criteria)
* Negative urine or serum pregnancy test on females of childbearing potential
* All females of childbearing potential and males must use an effective barrier method of contraception during the treatment period and for at least 1 month thereafter.

Exclusion Criteria:

* Chemotherapy or immunotherapy within 3 weeks of study entry
* Concomitant use of any other anti-cancer therapy
* Concomitant use of any other investigational agent
* Any known cardiac abnormalities such as:

  * Congenital long QT syndrome;
  * QTcF interval >480 milliseconds (msec);
  * A myocardial infarction within 12 months of study entry;
  * Other significant ECG abnormalities including 2nd atrio-ventricular (AV) block type II, 3rd degree AV block, or bradycardia (ventricular rate < 50 beats/ min).
  * An ECG recorded at screening showing significant ST depression (ST depression of ≥2 mm, measured from isoelectric line to the ST segment at a point 60 msec at the end of the QRS complex). If in any doubt, the patient should have a stress imaging study and, if abnormal, angiography to define whether or not CAD is present;
  * Congestive heart failure (CHF) that meets New York Heart Association (NYHA) Class II to IV definitions and/or ejection fraction <40% by MUGA scan or <50% by echocardiogram and/or MRI;
  * A known history of sustained ventricular tachycardia (VT), ventricular fibrillation (VF), Torsade de Pointes, or cardiac arrest unless currently addressed with an automatic implantable cardioverter defibrillator (AICD);
  * Hypertrophic cardiomyopathy or restrictive cardiomyopathy from prior treatment or other causes (if in doubt, see ejection fraction criteria above);
  * Any cardiac arrhythmia requiring anti-arrhythmic medication;
* Serum potassium <3.8 mmol/L or serum magnesium <0.85 mmol/L (electrolyte abnormalities can be corrected with supplementation to meet inclusion criteria)
* Concomitant use of drugs that may cause a prolongation of the QTcF
* Concomitant use of CYP3A4 inhibitors
* Impaired liver, renal or other organ function not caused by lymphoma, which will interfere with the treatment schedule
* Concomitant use of warfarin due to a potential drug interaction
* Clinically significant active infection
* Known infection with human immunodeficiency virus (HIV)
* Patient has known clinically active hepatitis B or C
* Previous extensive radiotherapy involving ≥30% of bone marrow (e.g., whole pelvis, half spine), excluding patients who have had total body irradiation as part of a conditioning regimen for stem cell transplant
* Major surgery within 2 weeks of study entry
* Peripheral neuropathy or neuropathic pain of Grade 2 or worse
* Platelet count <50 × 109 cells/L or platelet count <30 × 109 cells/L if bone marrow disease involvement is documented
* Serum creatinine >2.0 × ULN
* Patients who are pregnant or breast-feeding
* Patient has known hypersensitivity to any components of bortezomib (such as boron, mannitol), or panobinostat

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2009-11; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate | 1 year

SECONDARY OUTCOMES:
Time to response, Duration of response, Progression-free survival, Overall survival, Safety and tolerability, Changes in disease-related symptoms and ECOG performance status. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Yeow Tee Goh, MBBS MMed, Principal Investigator — Singapore General Hospital; Darryl Tan, MBBS MMED, Study Chair — Singapore General Hospital
Locations (5):
- Malaysia (2):
  - Hospital Universiti Kebangsaan Malaysia ( HUKM ), Kuala Lumpur, Kuala Lumpur
  - Subang Jaya Medical Centre, Subang Jaya, Selangor
- Singapore (2):
  - National Cancer Center, Singapore
  - Singapore General Hospital, Singapore
- Samsung Medical Centre, Seoul, Seoul, South Korea

REFERENCES:
- [Derived] Tan D, Phipps C, Hwang WY, Tan SY, Yeap CH, Chan YH, Tay K, Lim ST, Lee YS, Kumar SG, Ng SC, Fadilah S, Kim WS, Goh YT; SGH651 Investigators. Panobinostat in combination with bortezomib in patients with relapsed or refractory peripheral T-cell lymphoma: an open-label, multicentre phase 2 trial. Lancet Haematol. 2015 Aug;2(8):e326-33. doi: 10.1016/S2352-3026(15)00097-6. Epub 2015 Jul 7. PMID 26688485